CLINICAL TRIAL: NCT00535873
Title: A Phase II Study of Lenalidomide as Initial Treatment of Patients With Chronic Lymphocytic Leukemia Age 65 or Older.
Brief Title: Lenalidomide as Initial Treatment of Patients With Chronic Lymphocytic Leukemia (CLL) Age 65 and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0715
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Leukemia; CLL; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Leukemia; CLL; chronic lymphocytic leukemia; SLL; small lymphocytic lymphoma; Untreated CLL; Lenalidomide; CC-5013; Revlimid; Oral
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide starting dose of 5 mg (capsules) by mouth daily for 28 days, one cycle.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Starting dose of 5 mg (capsules) by mouth daily for 28 days, one cycle.
  Other Names: Revlimid; CC-5013

SUMMARY:
Primary Objective:

* To assess the activity of lenalidomide in patients with previously untreated chronic lymphocytic leukemia (CLL) age 65 and older.

Secondary Objective:

* To assess the tolerability of lenalidomide in patients with untreated CLL age 65 and older

DETAILED DESCRIPTION:
The Study Drug:

Lenalidomide is designed to change the body's immune system and may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Drug Administration:

If you are found to be eligible to take part in this study, you will take lenalidomide by mouth every morning at about the same time each day for 28 days. Twenty-eight (28) days is considered 1 cycle. The dose and schedule of lenalidomide may be adjusted up or down, depending on how the disease responds and the side effects you may experience. Swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

Concomitant Medications:

Allopurinol will be prescribed for you during the first 14 days of treatment. This medication is taken by mouth and will help protect your kidney function.

Study Visits:

During this study, you will have blood (about 1 tablespoon each) drawn every other week until the best dose of lenalidomide has been found. Blood tests (about 1 tablespoon each) may be done more often if the dose of medication needs to be changed or if you experience intolerable side effects. Women who are able to have children must have a negative urine or blood (less than 1 teaspoon) pregnancy test 10 - 14 days and 24 hours before starting lenalidomide therapy, even if they have not had a menstrual period due to treatment of the disease or had as little as one menstrual period in the past 24 months. If you have regular or no menstrual cycles, you will then have pregnancy tests every week for the first 4 weeks, then every 4 weeks while taking lenalidomide, again when you have been taken off of lenalidomide therapy, and then 28 days after you have stopped taking lenalidomide. If you have irregular menstrual cycles, you will have pregnancy tests every week for the first 4 weeks, then every 2 weeks while taking lenalidomide, again when you have been taken off of lenalidomide therapy, and then 14 days and 28 days after you have stopped taking lenalidomide. Every month for the first 3 months, then at Months 6, 9, 12, and 15 you will have a physical exam to see how you are doing. After the 15-month visit, you will have a physical exam every 6 months.

After the first 3 months, and then every 6 months after that (unless your study doctor does not think it is necessary), you will have a bone marrow biopsy and aspirate performed to check the status of the disease.

Length of Study:

You may stay on this study for as long as you are benefitting. You will be taken off this study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Lenalidomide is FDA approved and commercially available. Lenalidomide is approved for the treatment of patients with transfusion-dependent anemia due to Low- or Intermediate-1-risk myelodysplastic syndromes associated with the chromosome 5 abnormality with or without other chromosome abnormalities. Lenalidomide is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy. Its use in this study, for this disease, is investigational. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with untreated CLL or small lymphocytic lymphoma (SLL) with indication to treatment according to NCI Working Group guidelines.Patients that have received single agent rituximab will be allowed to participate in this study.
2. Age 65 or older
3. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0-2.
4. Adequate renal function indicated by serum creatinine less or equal to 2 and adequate hepatic function indicated as total bilirubin less or equal to upper level of normal and as alanine aminotransferase (ALT) less or equal 2 upper limit of normal (ULN).
5. Able to understand and sign Informed Consent after the investigational nature, study design, risks and benefits have been explained.
6. Able to adhere to the study visit schedule and other protocol requirements.
7. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation can be enrolled in the study as long as they have a reasonable expectation to have been cured with treatment modality received.
8. Females of childbearing potential (FCBP). A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence
9. Continued from above. from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing.
10. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy.
11. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
12. All patients must be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to Acetylsalicylic Acid (ASA) may use warfarin or low molecular weight heparin.

Exclusion Criteria:

1. Known sensitivity to thalidomide or its derivatives.
2. Documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood).
3. Known positivity for HIV or active hepatitis (B or C).
4. A serious medical condition, laboratory abnormality or psychiatric illness that would interfere with the ability of the patient to participate in this program according to the judgement of the Principal Investigator.
5. Active cardiovascular disease as defined by the New York Heart Association Class 3 or 4.
6. History of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Concurrent use of other chemotherapy agents.
8. Pregnant or breast feeding females. Lactating females must agree not to breast feed while taking lenalidomide.
9. No known history of tuberculosis or recent exposure to tuberculosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Takahashi K, Hu B, Wang F, Yan Y, Kim E, Vitale C, Patel KP, Strati P, Gumbs C, Little L, Tippen S, Song X, Zhang J, Jain N, Thompson P, Garcia-Manero G, Kantarjian H, Estrov Z, Do KA, Keating M, Burger JA, Wierda WG, Futreal PA, Ferrajoli A. Clinical implications of cancer gene mutations in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2018 Apr 19;131(16):1820-1832. doi: 10.1182/blood-2017-11-817296. Epub 2018 Jan 22. PMID 29358183
- [Derived] Strati P, Keating MJ, Wierda WG, Badoux XC, Calin S, Reuben JM, O'Brien S, Kornblau SM, Kantarjian HM, Gao H, Ferrajoli A. Lenalidomide induces long-lasting responses in elderly patients with chronic lymphocytic leukemia. Blood. 2013 Aug 1;122(5):734-7. doi: 10.1182/blood-2013-04-495341. Epub 2013 Jun 25. PMID 23801633
- [Derived] Badoux XC, Keating MJ, Wen S, Lee BN, Sivina M, Reuben J, Wierda WG, O'Brien SM, Faderl S, Kornblau SM, Burger JA, Ferrajoli A. Lenalidomide as initial therapy of elderly patients with chronic lymphocytic leukemia. Blood. 2011 Sep 29;118(13):3489-98. doi: 10.1182/blood-2011-03-339077. Epub 2011 Jul 1. PMID 21725050
- See also: M.D. Anderson Cancer Center's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 10/3/2007 through 7/10/2009. All participants recruited at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Sixty-one participants were registered and signed consent for this study. One participant signed consent but never received study medication.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One of the sixty-one participants who signed consent did not receive study medication and was not included in the analysis for this study.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 71 [66 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR defined as number of participants with best response of Complete Response (CR) or Partial Response (PR) out of total number of participants. CR is defined as absence of lymphadenopathy, hepatomegaly or splenomegaly on physical exam. Normal Complete Blood Count (CBC) with polymorphonuclear leukocytes >1500/µL, platelets >100,000/µL, hemoglobin >11.0 g/dL (untransfused); lymphocyte count <5,000/µL; Bone marrow aspirate and biopsy must be normocellular for age with <30% of nucleated cells being lymphocytes. Lymphoid nodules must be absent. PR requires a 50% decrease in peripheral lymphocyte count from , 50% reduction in lymphadenopathy, and/or 50% reduction in splenomegaly/hepatomegaly for a period of at least two months from completion of therapy. These patients must have one of the following: Polymorphonuclear leukocytes 1,500/µL or 50% improvement ; Platelets >100,000/µL or 50% improvement ; Hemoglobin >11.0 g/dL (untransfused) or 50% improvement from pre-treatment value.
Time Frame: From 3 cycles (90 days) up to 6 cycles (approximately 180 days)
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 60
participants | 39

ADVERSE EVENTS:
Time Frame: 5 years 4 months
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 24/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=60)
Anorexia (Gastrointestinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebrovascular Ischemia (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abnormal Coagulation tests (Blood and lymphatic system disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Fever (General disorders) | 4 (4)
Hernia Repair (Surgical and medical procedures) | 2 (2)
Hip Replacement Surgery (Surgical and medical procedures) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Necrosis (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Prostatic Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vessel injury lower extremity (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=60)
Fatigue (General disorders) | 32 (32)
Diarrhea (Gastrointestinal disorders) | 22 (22)
Tumor Flare (General disorders) | 16 (16)
Sencory Neuropathy (Nervous system disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 13 (13)
Constipation (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 10 (10)
Neurologic - Other (Nervous system disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Anorexia (Gastrointestinal disorders) | 9 (9)
Metabolic Laboratory abnormality (Metabolism and nutrition disorders) | 9 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Elevated Serum Creatinine (Metabolism and nutrition disorders) | 7 (7)
GI Pain (General disorders) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Peripheral Edema (Blood and lymphatic system disorders) | 6 (6)
Heartburn (Gastrointestinal disorders) | 6 (6)
Headache (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes